CLINICAL TRIAL: NCT07143006
Title: Innovative Application of Advanced Intelligent Electric Vehicles in Detecting and Analyzing Gait Abnormalities in Patients With Neurodegenerative Diseases, and Adding Value to the Creation of Improved Walking and Balance
Brief Title: Application of Smart Electric Vehicles in Analyzing Gait Abnormalities in Patients With Neurodegenerative Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Chien Tai Hong, Doctor, Professor, Principal Investigator, Taipei Medical University Shuang Ho Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: N202402036
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease; Dementia
Keywords: Neurodegenerative Diseases, Smart Electric Vehicles, Gait Training
MeSH Terms: conditions — Parkinson Disease; Dementia; Neurodegenerative Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Gait abnormalities in patients with neurodegenerative diseases.
  Interventions: Device: BestShape Go Intelligent Generation Transformable Electric Vehicle

INTERVENTIONS:
Device: BestShape Go Intelligent Generation Transformable Electric Vehicle — The specific applications of artificial intelligence in intelligent electric vehicles mainly include gait monitoring and analysis, real-time feedback and guidance, autonomous adaptive assistance, safety prevention and warnings, data collection and long-term tracking, as well as adding interactive and entertainment elements.

SUMMARY:
To explore the possibility of smart electric vehicles providing comprehensive gait assistance and improvement for patients with neurodegenerative diseases

DETAILED DESCRIPTION:
Background: Gait abnormalities are common in patients with neurodegenerative diseases, due to the disease's impact on the brain's ability to control movement coordination and balance, increasing the risk of falls and reducing the mobility of patients. There are no specific medications for treating these gait abnormalities. Non-pharmacological gait training is crucial in improving gait abnormalities in patients with neurodegenerative diseases. Gait training can bring significant benefits, such as improving walking ability and overall health and quality of life.

As Taiwan enters a super-aged society, the number of patients with neurodegenerative diseases is growing yearly. Despite Long-Term Care 2.0 addressing this issue, there is a lack of therapists, leading to insufficient training for patients. Therefore, an innovative way to promote gait training is needed. The use of Artificial Intelligence (AI)-driven smart electric vehicles for detecting and improving gait abnormalities is becoming feasible with the advancement of AI. This technology can monitor and analyze gait in real time and provide feedback to users to improve stride, speed, or balance. The application of AI smart electric vehicles in gait training and assistance for patients with neurodegenerative diseases could span multiple settings, including hospitals and subacute rehabilitation centers, residential care institutions, home environments, and community health centers and aging community hubs.

Inventec Medical Technology's BestShape Go Intelligent Generation Transformable Electric Vehicle represents profound care for the related population and those with mobility difficulties. This smart electric vehicle has dual modes of riding and assisted walking. The assisted walking function provides users with a sense of security and appropriate guidance while immediately tracking and detecting potential danger, making it a potential AI gait training partner.

Project Objective: To explore the possibility of smart electric vehicles providing comprehensive gait assistance and improvement for patients with neurodegenerative diseases. Research Design: As a phase one study, this project tests the ability of smart electric vehicles to detect and analyze the abnormal gait of patients with neurodegenerative diseases during short-term (60 minutes) gait training, and the improvement in walking and balance when using smart electric vehicles after training.

Research Goal: To assess the effect of detection and training under the guidance of smart electric vehicles in improving the walking speed and stability of patients with neurodegenerative diseases.

Research Method: The target group consists of patients diagnosed with mild neurodegenerative diseases and walking disabilities. Selection criteria include age, walking ability, cognitive status, etc. Inventec's smart vehicle is equipped with sensors for monitoring gait and analyzing gait data through AI. Participants undergo initial gait assessment, including walking speed and balance tests, using the 6-meter Timed-up-and-Go method. They then engage in 45 minutes of gait training, using the smart electric vehicle for stride adjustment, speed control, and balance practice, with real-time feedback. Finally, participants undergo the 6-meter Timed-up-and-Go test again to compare progress. Expected Outcome: Training with the smart electric vehicle will significantly improve the walking speed and balance ability of patients with neurodegenerative diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with neurodegenerative diseases(such as Parkinson's disease or dementia).
2. Age: 60-85 years.
3. Capable of walking to some extent, but may have mild to moderate gait disturbances.
4. Able to understand the trial procedures and give informed consent.

Exclusion Criteria:

1. Unable to walk or requiring comprehensive physical support.
2. Conditions such as heart disease, uncontrolled high blood pressure, or a history of major surgery.
3. Severe cognitive impairment preventing understanding of the trial procedures or giving informed consent.
4. Visual or auditory impairments severe enough to prevent following trial instructions.
5. Participation in other clinical trials within a certain period in the past, which could affect the assessment of results.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2025-08-20 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
6-meter Timed-up-and-Go method | 45 minutes of gait training

CONTACTS AND LOCATIONS:
Overall Officials: Lung Chan, MD, PhD, Principal Investigator — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Shuang Ho Hospital, New Taipei City, Taiwan